CLINICAL TRIAL: NCT07362134
Title: The Application of Point-by-point Pulsed-Field Ablation for Recurrent Atypical Flutter: Safety, Acute Success, Efficacy, and Outcome
Brief Title: Pulsed-Field Ablation for Recurrent Atypical Atrial Flutter
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-09-005C
Record Dates: First submitted 2025-12-23; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-12

CONDITIONS: Atypical Atrial Flutter; Atrial Flutter
Keywords: Atypical atrial flutter; Recurrent atrial flutter; Pulsed field ablation; Non-thermal catheter ablation; Catheter ablation; Electrophysiology study
MeSH Terms: conditions — Atrial Flutter

STUDY DESIGN:
Intervention Model Description: Single-center, prospective, non-randomized, single-arm study in which all enrolled subjects undergo catheter ablation with point-by-point pulsed-field ablation using the Biosense Webster Dual Energy system, with standardized electroanatomic mapping and protocol-driven follow-up including repeat electrophysiology study and imaging.
Masking Description: This is an open-label, single-arm study. All participants and investigators are aware of the treatment assignment, and no masking or blinding procedures are implemented.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Point-by-Point Pulsed-Field Ablation (PFA) (Experimental): All participants in this experimental arm will undergo catheter ablation for recurrent atypical atrial flutter using a point-by-point pulsed-field ablation strategy with the Biosense Webster Dual Energy system (TRUPULSE™ generator and Dual Energy THERMOCOOL SMARTTOUCH™ SF catheter) guided by CARTO™ 3 electroanatomic mapping. Linear or focal lesions will be created along the critical isthmus or scar-related circuit to achieve termination of atypical flutter and bidirectional conduction block. If bidirectional block cannot be achieved with pulsed-field ablation alone, radiofrequency energy using the same system may be applied as a bail-out at the operator's discretion.
  Interventions: Procedure: Point-by-point pulsed-field catheter ablation

INTERVENTIONS:
Procedure: Point-by-point pulsed-field catheter ablation — Point-by-point pulsed-field catheter ablation delivered with a dual-energy pulsed field/radiofrequency ablation system. The procedure is guided by 3D electroanatomic mapping to identify the critical isthmus or scar-related circuit responsible for recurrent atypical atrial flutter. Linear or focal lesions are created with point-by-point pulsed-field applications along the targeted line to achieve arrhythmia termination and durable bidirectional conduction block. Radiofrequency energy using the same catheter and generator may be applied only as a bail-out strategy if pulsed-field ablation alone fails to achieve the acute endpoint.

SUMMARY:
Recurrent atypical atrial flutter (AFL) after prior atrial fibrillation or flutter ablation remains challenging to treat, and conventional radiofrequency ablation may be limited by incomplete lesion formation and risk of collateral damage. Pulsed-field ablation (PFA) uses non-thermal electric fields to create myocardial lesions with relative sparing of surrounding tissues and may improve the safety and efficacy of ablation for atypical AFL.

This prospective, non-randomized, single-arm study will enroll approximately 30 patients with clinically documented recurrent atypical AFL who are referred for elective catheter ablation using a point-by-point pulsed-field ablation system. During the index procedure, detailed electroanatomic mapping will be performed to identify the critical isthmus or circuit, followed by linear or focal PFA and confirmation of bidirectional conduction block.

The primary safety endpoint is the incidence of procedure- and device-related primary adverse events. The primary effectiveness endpoint is acute procedural success, defined as termination of atypical AFL and establishment of bidirectional block across the targeted lesion set at the end of the procedure. Secondary endpoints include recurrence of any atrial arrhythmia during 12-month follow-up, durability of the linear lesions assessed by repeat electroanatomic mapping at 3 months, changes in atrial scar on cardiac MRI, peri-procedural changes in blood biomarkers, and the rate of serious adverse events related to the procedure or study device.

DETAILED DESCRIPTION:
Atypical atrial flutter (AFL) is a challenging atrial tachyarrhythmia that frequently occurs after prior catheter ablation for atrial fibrillation (AF) or AFL. Conventional radiofrequency ablation (RFA) can be limited by variable lesion size and depth, difficulty in achieving durable transmural linear block, and the risk of collateral injury to adjacent structures such as the esophagus, phrenic nerve, and coronary arteries. These limitations are particularly important in recurrent atypical AFL, where complex macro-reentrant or localized reentrant circuits often form along prior ablation scars or in regions of epicardial conduction in the posterior left atrium and pulmonary veins, making durable ablation difficult to achieve.

Pulsed-field ablation (PFA), based on non-thermal irreversible electroporation, has emerged as a promising technique that can create deep, contiguous lesions with preferential myocardial injury while sparing non-cardiac tissues. Early clinical experience with point-by-point PFA systems has demonstrated high acute and chronic success rates for pulmonary vein isolation and linear ablation with low complication rates in patients with recurrent AF or AFL after prior ablation. These data suggest that focal PFA may overcome some of the safety and efficacy limitations of conventional thermal energy sources.

This single-center, prospective, non-randomized, single-arm clinical investigation will enroll approximately 30 adult patients with clinically documented recurrent atypical AFL after prior AF/AFL ablation within 5 years who are scheduled for elective repeat ablation. The investigational system is the Biosense Webster Dual Energy Pulsed Field/Radiofrequency Ablation System, consisting of the TRUPULSE™ Generator, the Dual Energy THERMOCOOL SMARTTOUCH™ SF (STSF) catheter, and the CARTO™ 3 System with VISITAG SURPOINT™ Module. Standard-of-care adjunctive devices (e.g., OCTARAY™ mapping catheter, DECANAV™ diagnostic catheter, VIZIGO™ sheath, and intracardiac echocardiography [ICE] catheter) will be used as appropriate.

Eligible subjects are ≥18 years of age with recurrent atypical AFL documented by ECG or electrophysiologic study after prior pulmonary vein isolation and/or AFL ablation, including gap-reentrant, perimetral, roof-dependent, bi-atrial, or scar-related circuits, and who are willing and able to provide informed consent and complete follow-up. Key exclusion criteria include AFL due to reversible causes, recent major cardiac events or surgery, significant structural heart disease (e.g., severe valvular disease, hypertrophic cardiomyopathy, markedly enlarged left atrium), severe ventricular dysfunction, significant pulmonary or renal disease, active malignancy or infection, untreated severe sleep apnea, contraindication to anticoagulation, pregnancy, vulnerable populations, and limited life expectancy.

After signing informed consent, subjects will undergo baseline evaluations including 12-lead ECG, 14-day Holter monitoring, transthoracic echocardiography, transesophageal echocardiography, and cardiac MRI at least one day before the ablation procedure. Oral anticoagulation will be managed according to guideline-based practice, with at least 4 weeks of pre-procedural anticoagulation and continued post-procedural anticoagulation per current clinical standards.

The index procedure will be performed under general anesthesia or deep sedation. A deflectable decapolar catheter will be positioned in the coronary sinus. Double transseptal puncture will be performed under fluoroscopic and ICE guidance, followed by systemic heparinization to maintain an activated clotting time of 300-350 seconds. Bi-atrial electroanatomic maps will be created with the CARTO® 3 system and high-density mapping catheters. ICE will be used systematically for transseptal guidance, catheter navigation, and surveillance of pericardial effusion, posterior wall-esophagus distance, pulmonary vein ostial dimensions, and valvular function before, during, and after ablation. A transthoracic echocardiogram will be performed immediately after the procedure or before discharge to detect complications.

Mapping of atypical AFL or atrial tachycardia will follow established protocols from the investigators' prior work. If the patient is in sinus rhythm, arrhythmia will be induced using atrial pacing and isoproterenol infusion. High-density activation and entrainment mapping will be performed to characterize the reentrant circuit(s) or localized reentry, with post-pacing interval (PPI) analyses at multiple sites; a PPI within 20 ms of the tachycardia cycle length will be considered within the circuit. Circuits will be classified as macro-reentrant or localized reentry based on activation patterns.

Once the critical isthmus or focal source has been identified, the Dual Energy STSF catheter connected to the TRUPULSE™ Generator will be used to deliver point-by-point PFA along the targeted line of block or boundary of the critical zone, aiming to interrupt the reentrant loop or focal driver. Lesions will be applied at approximately 3-5 mm spacing with contact force maintained at 10-20 g. Pulse delivery and tag indices (PF Index/RF Tag Index) will be titrated according to anatomical location, with higher index targets at anterior sites and lower targets at posterior wall regions near the esophagus. A maximum number of applications per location will be predefined. The acute endpoint is termination and non-inducibility of atypical AFL and demonstration of bidirectional conduction block across any linear lesion, confirmed by activation mapping and differential pacing. If AFL does not terminate or bidirectional block cannot be achieved after up to two passes of PFA, conventional RFA using the same catheter and generator will be permitted as a bail-out strategy and considered acute treatment failure for the primary effectiveness endpoint.

After ablation, inducibility testing will be performed with burst atrial pacing, with or without isoproterenol, to confirm non-inducibility of atypical AFL. Peri-procedural complications and device-related events will be carefully monitored and recorded. Primary adverse events include major complications such as cardiac tamponade, stroke or transient ischemic attack, major vascular complications, atrioesophageal fistula, pulmonary vein stenosis, and procedure- or device-related death, among others, occurring within 7 days of the index ablation (or up to 90 days for delayed events as appropriate). Safety oversight will include pre-specified reporting to the sponsor, institutional review board, and regulatory authorities, as well as periodic review by an independent Data and Safety Monitoring Board (DSMB) with planned interim safety analyses.

All subjects will be followed clinically for 12 months after the index procedure. A 12-lead ECG will be obtained before hospital discharge. Outpatient follow-up visits will occur approximately 2 weeks after PFA and then every 1-3 months. At each visit, symptoms, medications, and adverse events will be assessed and ECGs recorded. Fourteen-day Holter monitoring will be scheduled at 3, 6, 9, and 12 months, and additional 24-hour Holter or event monitoring will be performed for symptomatic episodes. Recurrent AF/AFL is defined as any atrial tachyarrhythmia (AF, atrial tachycardia, or AFL) lasting >30 seconds after a 3-month blanking period.

Cardiac MRI with late gadolinium enhancement will be performed at baseline and at 3 and 12 months post-ablation to quantify atrial scar burden and evaluate changes in scar distribution and lesion durability over time. Blood biomarkers (including liver enzymes, cardiac enzymes, inflammatory markers, and haptoglobin) will be collected before and after ablation and at 3, 6, 9, and 12 months to characterize myocardial injury and inflammatory responses to dual-energy ablation.

All patients will be recommended to undergo a repeat electrophysiology study and repeat electroanatomic mapping at approximately 3 months (±4 weeks) to directly assess the durability of PFA linear lesions and confirm persistent bidirectional block across prior ablation lines. In cases of reconnection of previous PFA lines, touch-up RFA will be performed per investigator discretion. However, reconnection without documented atrial arrhythmia lasting >30 seconds will not count as a clinical recurrence for the secondary effectiveness endpoint.

The primary safety endpoint is the incidence of predefined primary adverse events within 7 days of the index procedure. The primary effectiveness endpoint is acute procedural success, defined as termination and non-inducibility of atypical AFL with confirmed bidirectional block across ablation lines at the end of the procedure. Secondary endpoints include freedom from recurrent atrial arrhythmias at 12 months, durability of linear lesions on repeat mapping, changes in atrial scar on MRI, serial biomarker profiles, and serious adverse events related to the procedure and/or investigational device.

This feasibility study is designed to generate prospective clinical data on the safety, acute procedural success, arrhythmia outcomes, lesion durability, and myocardial/inflammatory response associated with point-by-point PFA using the BWI Dual Energy system in patients with recurrent atypical AFL after prior ablation. The results are expected to inform future larger studies and may help refine ablation strategies and energy delivery parameters for complex post-ablation atrial tachyarrhythmias.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clinically documented recurrent atypical AFL (based on ECG findings or electrophysiological study findings) after previous ablation for pulmonary vein isolation or atypical AFL within 5 years. The use of oral anticoagulation will follow current guidelines before and after the ablation procedure. In brief, oral anticoagulation will be administered for at least 4 weeks before the procedure.
2. Patients undergoing elective AFL ablation using point-by-point PFA (BWI PFA/RFA ablation system), for any of the following types of atypical AFL: gap reentrant, perimetral, roof-dependent, bi-atrial, or scar-related atypical AFL.
3. Patients aged ≥18 and <80.
4. Patient is willing and capable of providing informed consent.
5. Patient is willing and capable of participating in all follow-up assessments and testing associated with this clinical investigation at an approved clinical investigation center.

Exclusion Criteria:

1. those with AFL due to reversible conditions (e.g., thyroid disorders, acute alcohol intoxication, or recent major surgeries),
2. those who had acute coronary syndrome, underwent percutaneous coronary intervention, or had valve or coronary bypass grafting surgery in the 90 days preceding the procedure, or receiving surgical interventions with mechanical valve implants, and
3. those with documented cardiac thrombus before the procedure, a history of cardiac thrombus, stroke, or transient ischemic attack in the previous 90 days.
4. Categorized as vulnerable population and requires special treatment with respect to safeguards of well being.
5. Any of the following atrial conditions:

   1. Left atrial anteroposterior diameter ≥ 5.5 cm, or if LA diameter not available, non-indexed volume >100 ml (physician note or imaging)
   2. Current atrial myxoma
   3. Any PV abnormality, stenosis, or stenting (common and middle PVs are admissible)
6. Any of the following CV conditions:

   1. History of sustained ventricular tachycardia or any ventricular fibrillation
   2. Current or anticipated pacemaker, implantable cardioverter defibrillator or cardiac resynchronization therapy devices, or implantable loop recorder.
   3. Prior interatrial baffle, atrial septal patch, atrial septal defect closure device, patent foramen ovale occluder, Amulet devices, or other left atrial appendage closure device if implanted within 90 days of enrollment
7. Presence of any of the following:

   1. Moderate to severe mitral valve stenosis
   2. More than moderate mitral regurgitation (>3+)；
   3. Moderate to severe aortic stenosis
8. Hypertrophic cardiomyopathy
9. Any IVC filter, known inability to obtain vascular access or other contraindication to femoral access
10. Awaiting cardiac transplantation or other cardiac surgery within the next 12 months
11. Severe right ventricular dysfunction with documented echocardiography and/or hemodynamic data within 6 months.
12. Any of the following conditions at baseline:

    1. Heart failure associated with NYHA Class III or IV
    2. Documented LVEF < 40% as documented within the previous 12 months
    3. Any of the following events within 90 Days of the Consent Date:

    i. Heart failure hospitalization: Heart failure hospitalization ii. Pericardium: Pericarditis or symptomatic pericardial effusion iii. GI bleeding: Gastrointestinal bleeding iv. Neurovascular event: Stroke, TIA, or intracranial bleeding v. Thromboembolism: Any active non-neurologic thrombus and/or thromboembolic event vi. Carotid intervention: Carotid stenting or endarterectomy vii. Diabetes: Uncontrolled diabetes mellitus or a recorded HgbA1c > 8.0%
13. Any of the following congenital conditions:

    1. Congenital heart disease: Congenital heart disease with any clinically significant residual anatomic or conduction abnormality
    2. Methemoglobinemia: History of known congenital methemoglobinemia
    3. G6PD deficiency: History of known G6PD deficiency
14. Any of the following known pre-existing conditions:

    1. Transplantation: Solid organ or hematologic transplant, or currently being evaluated for a transplant
    2. Diaphragmatic abnormality: Any prior history or current evidence of hemi-diaphragmatic paralysis or paresis
    3. Pulmonary: Severe lung disease, severe pulmonary hypertension, or any lung disease involving abnormal blood gases or requiring supplemental oxygen
    4. Renal: Renal insufficiency if an estimated glomerular filtration rate (eGFR) is < 30 mL / min / 1.73 m2, or with any history of renal dialysis or renal transplant
    5. Malignancy: Active malignancy at enrolment (other than squamous cell carcinoma)
    6. Gastrointestinal: Clinically significant gastrointestinal problems involving the esophagus or stomach including severe or erosive esophagitis, uncontrolled gastric reflux, gastroparesis, esophageal candidiasis or active gastroduodenal ulceration
    7. Infections: Active systemic infection
    8. Sleep apnea: Untreated diagnosed obstructive sleep apnea with apnea hypopnea index classification of severe (>30 pauses per hour)
    9. Hematologic condition: Known coagulopathy or bleeding disorder (e.g. von Willebrand disease, hemophilia)
    10. Contraindication to anticoagulation: Contraindication to, or unwillingness to use, systemic anticoagulation, or acceptable alternatives, pre-, intra- and post-procedure to achieve adequate anticoagulation.
    11. Pregnancy: Women of childbearing potential who are pregnant, lactating, not using medical birth control or who are planning to become pregnant during the anticipated study period
    12. General health conditions: Health conditions that in the investigator's medical opinion would prevent participation in the study, interfere with assessment or therapy, significantly raise the risk of study participation, or modify outcome data or its interpretation.
    13. Participation in another trial: Subjects who are currently enrolled in another investigational study or registry that would directly interfere with the current study, except when the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments; each instance must be brought to the attention of the Sponsor to determine eligibility.
    14. Life expectancy: Predicted life expectancy less than three years
15. A subject that is ineligible for participation for any other reason as determined by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of primary adverse events within 7 days of the index ablation procedure | Within 7 days after the index ablation procedure
  Proportion of subjects experiencing one or more predefined primary adverse events (PAEs) related to the procedure and/or investigational dual-energy ablation system within 7 days after the index ablation procedure. PAEs include major complications such as cardiac tamponade, stroke or transient ischemic attack, major vascular complications, atrioesophageal injury, pulmonary vein stenosis, and procedure- or device-related death, as defined in the protocol.
Acute procedural success of atypical atrial flutter ablation | At the end of the index ablation procedure
  Proportion of subjects in whom acute procedural success is achieved at the end of the index ablation procedure. Acute procedural success is defined as termination and non-inducibility of the clinical atypical atrial flutter and achievement of bidirectional conduction block across the targeted ablation line, confirmed by differential pacing. Cases requiring additional radiofrequency ablation because pulsed-field ablation alone cannot terminate the arrhythmia or achieve bidirectional block will be classified as acute treatment failures.

SECONDARY OUTCOMES:
Freedom from recurrent atrial arrhythmias | From the end of the 3-month blanking period through 12 months after the index ablation procedure.
  Proportion of subjects who are free from any documented atrial arrhythmia, including atrial fibrillation, atrial flutter, or atrial tachycardia, lasting > 30 seconds during follow-up after a 3-month blanking period following the index ablation procedure.

OTHER OUTCOMES:
Durability of pulsed-field linear lesions on repeat electroanatomic mapping | Approximately 3 months (± 4 weeks) after the index ablation procedure.
  Proportion of pulsed-field ablation linear lesions that remain electrically intact, with confirmed bidirectional conduction block across the ablation line, on repeat electroanatomic mapping during a planned repeat electrophysiology study.
Change in left atrial scar burden on cardiac MRI with late gadolinium enhancement | Baseline, 3 months, and 12 months after the index ablation procedure.
  Change in the extent of left atrial scar, expressed as the percentage of left atrial wall volume demonstrating late gadolinium enhancement on cardiac MRI, between baseline and follow-up scans after ablation.
Serial changes in serum cardiac troponin I/T levels | Baseline, within 24 hours after the index ablation procedure, and at 3, 6, 9, and 12 months after the index ablation procedure.
  Time course and magnitude of changes in serum cardiac troponin I or T levels as a biomarker of myocardial injury before and after ablation and during follow-up.
Serial changes in serum creatine kinase (CK) and CK-MB levels | Baseline, within 24 hours after the index ablation procedure, and at 3, 6, 9, and 12 months after the index ablation procedure.
  Time course and magnitude of changes in serum creatine kinase (total CK) and CK-MB levels as biomarkers of myocardial injury before and after ablation and during follow-up.
Serial changes in serum myoglobin levels | Baseline, within 24 hours after the index ablation procedure, and at 3, 6, 9, and 12 months after the index ablation procedure.
  Time course and magnitude of changes in serum myoglobin levels as an early biomarker of muscle and myocardial injury before and after ablation and during follow-up.
Serial changes in serum lactate dehydrogenase (LDH) levels | Baseline, within 24 hours after the index ablation procedure, and at 3, 6, 9, and 12 months after the index ablation procedure.
  Time course and magnitude of changes in serum lactate dehydrogenase levels as a marker of tissue injury before and after ablation and during follow-up.
Serial changes in serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels | Baseline, within 24 hours after the index ablation procedure, and at 3, 6, 9, and 12 months after the index ablation procedure.
  Time course and magnitude of changes in serum ALT and AST levels to assess systemic tissue injury and potential extracardiac effects before and after ablation and during follow-up.
Serial changes in systemic inflammatory biomarkers | Baseline, within 24 hours after the index ablation procedure, and at 3, 6, 9, and 12 months after the index ablation procedure.
  Time course and magnitude of changes in systemic inflammatory biomarkers, including C-reactive protein (CRP) , before and after ablation and during follow-up.
Serial changes in systemic inflammatory biomarker - erythrocyte sedimentation rate (ESR) | Baseline, within 24 hours after the index ablation procedure, and at 3, 6, 9, and 12 months after the index ablation procedure.
  Time course and magnitude of changes in systemic inflammatory biomarkers, including erythrocyte sedimentation rate (ESR), before and after ablation and during follow-up.
Serial changes in hemolysis-related biomarkers | Baseline, within 24 hours after the index ablation procedure, and at 3, 6, 9, and 12 months after the index ablation procedure.
  Time course and magnitude of changes in serum haptoglobin levels as a biomarker of hemolysis before and after ablation and during follow-up.
Serious adverse events related to the procedure and/or study device through 12 months | Up to 12 months after the index ablation procedure.
  Incidence of serious adverse events considered related to the catheter ablation procedure and/or the investigational dual-energy pulsed-field/radiofrequency ablation system during follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the current study protocol and informed consent do not include provisions for external IPD sharing, and the dataset contains detailed clinical, imaging, and electrophysiologic information that may pose a risk of re-identification. Study findings will be disseminated in aggregate form through scientific publications and presentations.